CLINICAL TRIAL: NCT05798598
Title: Evaluation of the Acquisition of Competencies and Participants' Satisfaction After a Scientific Writing Course: Comparison of Face-to-face and Online Modalities Through a Non-randomized Open Clinical Trial (SCRIU-B Study)
Brief Title: Evaluation of Competencies in Scientific Writing and Attendees' Satisfaction After Two Different Types of Training Courses: SCRIU-B Study
Acronym: SCRIU-B
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Dr. Antoni Esteve Foundation (Other)
Collaborators: Institut Català d'Oncologia (Other); University of Barcelona (Other); Ciber de Enfermedades Respiratorias (Unknown); University of Valencia (Other); CIBER de Epidemiología y Salud Pública (Unknown); University of Alicante (Other); Institut d'Investigació Biomèdica de Bellvitge (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: FDAE20220714
Record Dates: First submitted 2022-09-21; First posted 2023-04-04 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: Scientific Writing Training Course
Keywords: clinical trial design; continuing medical education; experimental design; medical writing; publishing; personal satisfaction
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Intervention Model Description: Non-randomized trial type
Masking Description: No masking. Each participant knows which group they belong to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- GIP - Face-to-face intervention group (Active Comparator): Participants in the scientific writing face-to-face training course.
  Interventions: Other: Scientific writing training course
- GIO: Online intervention group (Active Comparator): Participants in the scientific writing online training course.
  Interventions: Other: Scientific writing training course
- GIC: Control intervention group (No Intervention): Participants in other face-to-face training courses not related to scientific writing.

INTERVENTIONS:
Other: Scientific writing training course — Attendance to a training course on scientific writing. Attendees learn about the importance of scientific writing, structure and writing an original paper, how scientific publishing works, as well as how to interact with journal editors and reviewers.
  Arms: GIO: Online intervention group; GIP - Face-to-face intervention group

SUMMARY:
Scientific writing is one of the competencies required and requested by health professionals. There are several course formats designed for acquiring these competencies, although the improvement after taking part in these courses is not always demonstrated. Through an open and non-randomized experimental design, the SCRIU-B study aims to evaluate the acquisition of competencies in scientific writing after specific training courses (face-to-face and online) as well as the satisfaction of the participants with these courses. A control group with participants from other training workshops not related to scientific writing is included. Through different questionnaires about knowledge, attitudes, and skills we will evaluate and compare the improvement of their scientific writing skills. The results of the study will allow us to assess the usefulness of these courses and improve their format and implementation.

DETAILED DESCRIPTION:
Scientific writing and scientific publications are fundamental to the advancement of science in general. However many science degrees do not have specific writing courses. Several initiatives have attempted to improve scientific writing skills through face-to-face or online courses. However, few studies have analyzed the short- and long-term outcomes of these training interventions. Our objective is to evaluate the short- and long-term skills in scientific writing and the level of satisfaction of a group of students after taking a scientific writing course, in two training modalities (face-to-face and online).

The study will assess the scientific writing skills of those attending the course "Cómo redactar un artículo científico" in face-to-face and online format during 2019 and 2022 through a non-randomized open trial type study with a comparison group. The study will use questionnaires to analyze the participants' satisfaction with the course, their knowledge about scientific writing, and their attitude and skills toward scientific writing (knowledge, attitudes, and skills). The satisfaction questionnaire will be provided immediately after the course. The scientific writing skills of the attendees will be compared with a control group. The study is estimated to analyze the results of 270 participants, 90 per group. This protocol has been reviewed and approved by an ethics committee.

The study will be carried out between 2019 and 2022 and participants will be recruited from 6 face-to-face and 4 online editions of the scientific writing course. We aim to analyze the real impact these seminars have on the scientific writing skills of their participants and demonstrate that face-to-face courses are more useful than online courses.

ELIGIBILITY:
Inclusion Criteria:

* Participants of the Esteve Foundation training workshops

Exclusion Criteria:

* Students who do not accept to participate in the study at the time of enrolment for the training course.
* Students who attended/enrolled in a Esteve Foundation's scientific writing course (face-to-face or online) prior to the study.
* Students who enroll in another Esteve Foundation's scientific writing course during the duration of the study.
* Students who have enrolled in other courses on scientific writing 12 months prior to recruitment for this study or during the duration of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2019-07-05 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Participants' satisfaction about the training course | 2 to 62 days
  Participants' satisfaction will be collected through a 14-item opinion questionnaire about the course with a Likert scale from 0 (minimum) to 10 (maximum). These 14 items include: overall opinion of the course, usefulness of the materials, usefulness of the in-class exercises, teaching capacity of the lecturers, duration of the course, usefulness of the new knowledge acquired in their current job, etc. Data will be analyzed using descriptive statistics. Items and overall scores will be compared between each of the 3 groups/arms of the study.
Participants' knowledge about scientific writing | 20 months
  Participants' general knowledge about scientific writing will be analyzed through a multiple-choice 8-item test that each participant will have to answer three times throughout the study (before, after and 18 months after the intervention). The knowledge test includes specific questions about scientific style, authorship requirements, editorial policies and characteristics of an original scientific article, among others. Correct answers will score 1 point and incorrect answers will score 0 (zero) points. Increase or decrease in knowledge will be determined by the differences through time in the overall scores of the three groups/arms of the study, differences on overall scores by participant (whole test) and differences by item and participant (score differences of the same item through time of the same participant). Data will be analyzed using descriptive statistics. Items and overall scores will be compared between each of the 3 groups/arms of the study.
Participants' attitudes towards scientific writing | 20 months
  Participants' opinion about their own capability towards scientific writing will be analyzed through a 5-item capability questionnaire with a Likert scale from 0 (minimum, not capable at all) to 10 (maximum, completely capable). The participants will state their opinion on their personal capability to write different types of scientific texts related to the publication of a scientific article such as scientific manuscripts for national and international audiences, abstracts, the presentation letter and the answers to the reviewers. Increase or decrease in capability will be determined by differences through time in the overall scores for each participant (whole test), overall score by group/arm and differences by item and participant through time. Data will be analyzed using descriptive statistics. Items and overall scores will be compared between each of the 3 groups/arms of the study.
Students' skills in scientific writing | 20 months
  Participants' skills in scientific writing will be analyzed by comparing the number and types of scientific publications and their authorship role in them before and 18 months after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Felix Bosch, MD PhD, Study Director — Director
Locations (1):
- Dr. Antoni Esteve Foundation, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Seres E, Fernandez E, Garcia AM, Vives-Cases C, Bosch F. [Evaluation of competences in scientific writing after two different types of training courses: SCRIU-B study protocol]. Gac Sanit. 2022 Mar-Apr;36(2):188-192. doi: 10.1016/j.gaceta.2020.12.036. Epub 2021 Apr 15. Spanish. PMID 33865630